CLINICAL TRIAL: NCT03627611
Title: A Randomized Crossover Study, Examining Differential Effects of Levothyroxine and Liothyronine
Brief Title: Identification of Non-responders to Levothyroxine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Hormonlaboratoriet (Unknown); Spesialistsenteret Pilestredet Park (Unknown)
Responsible Party: Principal Investigator, Erik Fink Eriksen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/1883 (REK); 2017-003673-34 (EudraCT Number)
Record Dates: First submitted 2018-05-25; First posted 2018-08-13 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hypothyroidism; Biomarkers; Endocrine System Diseases
Keywords: Thyroxine; Triiodothyronine
MeSH Terms: conditions — Hypothyroidism; Endocrine System Diseases | interventions — Thyroxine; Triiodothyronine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T4 (Active Comparator)
  Interventions: Drug: Levothyroxin
- T3 (Experimental)
  Interventions: Drug: Liothyronine

INTERVENTIONS:
Drug: Levothyroxin — 3 months
  Arms: T4
Drug: Liothyronine — 3 months
  Arms: T3

SUMMARY:
The purpose of this study is to assess differential effects of T4 and T3 on cell and tissue level

DETAILED DESCRIPTION:
15-20% of the patients with hypothyroidism remain symptomatic, despite adequate thyroxine substitution. Endocrinologists are split in their opinion on combination therapy with T4 and T3 on patients with poorly regulated hypothyroidism. There are no objective means, by which to identify individuals who would benefit from combination therapy. The purpose of this study is to assess differential effects of T4 and T3 on body temperature, metabolism, muscle strength and brain function. The main aim is to try to identify biomarkers reflecting different effects of T4 and T3 on cell and tissue level.

ELIGIBILITY:
Inclusion Criteria:

* Poorly regulated hypothyroidism
* Female aged between 18 and 65 years
* Written informed consent obtained from the patient according to national regulations

Exclusion Criteria:

* Cardiovascular disease
* Chronic liver disease
* Chronic kidney disease
* Any other endocrinological disease
* Use of beta blockers
* Pregnant or lactating females
* Hormonal substitution other than T3 and T4
* Known psychiatric disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 69 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Brown adipose tissue activation | 6 months
  Thermal imaging of supraclavicular fossa

SECONDARY OUTCOMES:
Body temperature | 6 months
  Rectal thermometer
Energy expenditure | 6 months
  Indirect calorimetry
Muscle strength | 6 months
  Hand grip test
ThyPRO Questionnaire | 6 months
  Thyroid patient reported outcome, 13 multi-item scale, range 0-100 with higher scores indicating poorer health status
Mean levels of thyroid hormones | 6 months
  TSH, free T4 and free T3
SF-36 Questionnaire | 6 months
  Short form health survey, 8 multi-item scale, range 0-100 with higher scores indicating better health status
Fatigue Questionnaire | 6 months
  11 item, range 0-33 with higher scores implying higher levels of fatigue
New biomarkers | 6 months
  Bone marrow fat, serum and urine
Micro-RNA, miR-92a | 6 months
  Serum exosomes

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fink Eriksen, Professor, Principal Investigator — Department of Endocrinology, Morbid Obesity and Preventive Medicine
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Bjerkreim BA, Hammerstad SS, Gulseth HL, Berg TJ, Lee-Odegard S, Eriksen EF. Thyroid Signaling Biomarkers in Female Symptomatic Hypothyroid Patients on Liothyronine versus Levothyroxine Monotherapy: A Randomized Crossover Trial. J Thyroid Res. 2022 May 4;2022:6423023. doi: 10.1155/2022/6423023. eCollection 2022. PMID 35572853
- [Derived] Bjerkreim BA, Hammerstad SS, Gulseth HL, Berg TJ, Omdal LJ, Lee-Odegard S, Eriksen EF. Effect of Liothyronine Treatment on Quality of Life in Female Hypothyroid Patients With Residual Symptoms on Levothyroxine Therapy: A Randomized Crossover Study. Front Endocrinol (Lausanne). 2022 Feb 22;13:816566. doi: 10.3389/fendo.2022.816566. eCollection 2022. PMID 35273566
- [Derived] Bjerkreim BA, Hammerstad SS, Gulseth HL, Berg TJ, Lee-Odegard S, Rangberg A, Jonassen CM, Budge H, Morris D, Law J, Symonds M, Eriksen EF. Effect of Liothyronine Treatment on Dermal Temperature and Activation of Brown Adipose Tissue in Female Hypothyroid Patients: A Randomized Crossover Study. Front Endocrinol (Lausanne). 2021 Nov 19;12:785175. doi: 10.3389/fendo.2021.785175. eCollection 2021. PMID 34867829